CLINICAL TRIAL: NCT00803699
Title: Predicting Dietary Selenium Needs to Achieve Target Blood Selenium Levels
Acronym: LoDoSe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GFHNRC009; NCI Agreement#Y1-CN-2017-04
Record Dates: First submitted 2008-12-03; First posted 2008-12-05 (Estimated); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Nutritional Requirements
Keywords: selenium
MeSH Terms: interventions — Selenium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Capsule contains no selenium
  Interventions: Dietary Supplement: placebo
- Selenium as L-selenomethionine (Active Comparator): 50, 100, or 200 micrograms of selenium
  Interventions: Dietary Supplement: selenium as L-selenomethionine

INTERVENTIONS:
Dietary Supplement: placebo — daily placebo capsules for 12 months
  Arms: Placebo
Dietary Supplement: selenium as L-selenomethionine — daily capsules of 50, 100, or 200 micrograms of L-selenomethionine for 12 months
  Arms: Selenium as L-selenomethionine

SUMMARY:
In this study, we will evaluate the effectiveness of several doses of oral selenomethionine in raising biomarkers of selenium status including plasma selenium concentrations.

DETAILED DESCRIPTION:
Results of studies with animal tumor models and human clinical trials suggest that the essential nutrient selenium can be anti-tumorigenic if consumed at levels greater than nutritional requirements. If it is possible to increase plasma selenium concentrations above 120 nanograms per milliliter with less than 200 micrograms of selenium daily, then it is possible that supplementation can be accomplished through the use of selenium-containing foods.

ELIGIBILITY:
Inclusion Criteria:

* able to swallow capsules
* body mass index less than 40

Exclusion Criteria:

* Pregnancy
* Chronic liver or kidney disease
* taking medication that might affect liver and/or kidney
* blood pressure 140/90 or higher
* already taking more than 50 micrograms of selenium

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2005-11; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of effectiveness of consuming oral doses of L-selenomethionine in raising plasma selenium concentrations | Baseline, and after 3, 6, 9, and 12 months of supplementation

SECONDARY OUTCOMES:
Biomarkers of selenium status will be determined in urine, buccal cells, and plasma. White blood cells will be analyzed to identify DNA damage, reflecting the degree of oxidative damage and evaluate the status of antioxidant repair mechanisms. | Baseline and after 12 months of supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Gerald F Combs, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

REFERENCES:
- [Background] Jackson MI, Combs GF Jr. Selenium and anticarcinogenesis: underlying mechanisms. Curr Opin Clin Nutr Metab Care. 2008 Nov;11(6):718-26. doi: 10.1097/MCO.0b013e3283139674. PMID 18827575